CLINICAL TRIAL: NCT05766540
Title: Effect of add-on Aripiprazole on Cardiometabolic Profile in Treatment Resistant Schizophrenia With Metabolic Syndrome: A Randomized Controlled Trial
Brief Title: Add-on Aripiprazole on Cardiometabolic Profile in Treatment Resistant Schizophrenia: RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Debadatta Mohapatra, Assistant Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T/IM-F/21-22/30
Record Dates: First submitted 2023-02-17; First posted 2023-03-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Difference in the Change in Cardiovascular Risk in Treatment Resistant Schizophrenia
MeSH Terms: interventions — Aripiprazole; Clozapine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aripiprazole (Experimental): This group will receive Aripiprazole 10 mg/day for 6 months along with Clozapine and Metformin
  Interventions: Drug: Aripiprazole 10 MG
- Treatment as usual (Placebo Comparator): This group will receive Clozapine and Metformin.
  Interventions: Drug: Aripiprazole 10 MG

INTERVENTIONS:
Drug: Aripiprazole 10 MG — Aripiprazole hroup will receive Aripiprazole 10 mg/day along with Clozapine and Metformin
  Other Names: Clozapine, Metformin 1000 mg

SUMMARY:
The goal of this clinical trial participant population is to evaluate the effect of add on Aripiprazole in reducing the metabolic parameters in patients of TRS on Clozapine with metabolic syndrome. The cardiovascular risk would be measured by calculating the change in QRISK3(QRISK3 is an algorithm tool used to calculate cardiovascular risk. The software calculates the risk score using various parameters. It is a name not an abbreviation.) score and the metabolic parameters by change in Low density lipoprotein(LDL)/High-density lipoprotein(HDL) ratio, High sensitive C Reactive Protein (hs CRP), Insulin resistance (HOMA IR) and fasting plasma glucose level. The main question is to find out the change in cardiovascular risk score between the study groups in TRS on Clozapine with metabolic syndrome. It aims to answer the change in cardiovascular risk in terms of change in QRISK 3 score.

* Participants will be assessed for cardiovascular risk using QRISK 3 and entering the entering information like age, height, BMI, weight, Lipid profile, past history of angina, Chronic Kidney Disease (CKD), Migraine etc in the QRISK 3 algorithm.
* Subsequently they will be assessed using rating scales like Positive and negative symptom scale (PANSS) and Clinical Global Improvement (CGI) for positive and negative symptoms and clinical global improvement respectively.
* They will be randomized into 2 groups and one group will receive treatment as usual while the other group will receive Aripiprazole 10 mg/day along with treatment as usual.
* They will be reassessed at 3 time points like baseline, at 3 months and 6 months.
* Blood sample will be collected for hs CRP, lipid profile, Fasting Blood Sugar (FBS) at the baseline and after 6 months.

Researchers will compare both the groups to see if augmentation with Aripiprazole will reduce the metabolic risk or not.

DETAILED DESCRIPTION:
Schizophrenia (SCZ) is a chronic severe mental illness usually having an unremitting course and associated with gross socio occupational deterioration. Patients of SCZ and other severe mental illness experience higher prevalence of physical morbidity like cardiovascular diseases, weight gain, obesity, dyslipidaemia, diabetes mellitus and metabolic syndrome as compared to general population. Life expectancy of patients with SCZ is reduced by approximately 20 years than general population because of cardiovascular morbidities. In patients with SCZ, data suggests that 1 in every 3 patients have metabolic syndrome, 1 in every 2 patients are overweight, 1 in 5 have significant hyperglycaemia and 2 in every 5 patients have dyslipidaemia. Atypical antipsychotics like Olanzapine and Clozapine used to treat patients of SCZ have highest association with obesity, metabolic syndrome and other cardiovascular complications. Significant percentage (25%) of patients with SCZ tends to show poor response to antipsychotics, eventually requiring Clozapine treatment. Clozapine is the only US FDA approved treatment for treatment resistant schizophrenia (TRS), but around 28-45% of patients on long term Clozapine use eventually tend to develop metabolic syndrome during the treatment course. Hence, there is a need to search for drugs which can be used in combination with Clozapine for the treatment of Clozapine induced metabolic syndrome. Metformin, an oral hypoglycaemic agent has been a recommended treatment for type 2 diabetes mellitus and also for antipsychotic induced metabolic syndrome. In a metanalysis of 4 RCTs on TRS patients on Clozapine with metabolic syndrome, it has been found that add-on Metformin is consistently found to have superior efficacy over placebo in reducing metabolic syndrome. However, metformin use causes subclinical lactic acidosis and hence it's use has been discouraged in patients with hepatic impairment, heart failure and chronic kidney disease as it requires close monitoring of renal function test and serum B12. The exact duration of metformin treatment for antipsychotic induced metabolic syndrome has been inconsistent. Hence, there is a need for searching alternative which can reduce Clozapine associated metabolic side effects along with beneficial effects on psychopathology in treatment resistant scenarios. Aripiprazole, a partial D2 agonist and post synaptic D2 antagonist is used as a successful augmenting agent in TRS. In patients with schizophrenia with metabolic syndrome, add-on Aripiprazole has been found to be superior to placebo in reducing metabolic syndrome in a metanalysis of 4 RCTs. They have measured biochemical parameters like CRP, Insulin resistance (HOMA IR), LDL/TG ratio as outcome measures to substantiate their findings.

In this study the investigators would like to evaluate the effect of add on Aripiprazole in reducing the metabolic parameters in patients of TRS on Clozapine with metabolic syndrome. In our study the investigators would measure the cardiovascular risk by calculating the change in QRISK3 score and the metabolic parameters by change in LDL/HDL ratio, hs CRP, Insulin resistance (HOMA IR) and fasting plasma glucose level.

3.RESEARCH HYPOTHESIS: Null hypothesis: There will be no significant difference in the change in cardiovascular risk score between the study groups in TRS on Clozapine with metabolic syndrome.

Alternative hypothesis: There will be significant difference in the change in cardiovascular risk score between the study groups in TRS on Clozapine with metabolic syndrome.

4. OBJECTIVES: Primary

1. To evaluate the effect of add-on Aripiprazole on Cardiometabolic profile in terms of change in Q RISK 3 score over a period of 6 months in patients with TRS on Clozapine with Metabolic syndrome.

Secondary

1. To evaluate the effect add-on Aripiprazole in terms of the change in LDL/HDL ratio over a period of 6 months in patients with TRS on Clozapine with Metabolic syndrome.
2. To evaluate the effect of add-on Aripiprazole versus Metformin on insulin resistance (HOMA IR) over a period of 6 months in patients with TRS on Clozapine with Metabolic syndrome.
3. To evaluate the effect of add-on Aripiprazole versus Metformin on hs-CRP over a period of 6 months in patients with TRS on Clozapine with Metabolic syndrome
4. To evaluate the safety of Clozapine, Aripiprazole and Metformin in terms of reported adverse events.

METHODOLOGY:

Study Population & Eligibility The study population will comprise of 60 patients with TRS (TRRIP consensus criteria) on Clozapine monotherapy, attending the in-patient or out-patient department of Psychiatry, All India Institute of Medical Sciences, Bhubaneswar.

Tools to be used:

1. QRISK3 2018 algorithm - it is used to calculate the cardiovascular risk in the upcoming 10 years. The risk is calculated for participants between the age group of 25 to 84 years after entering information like age, height, BMI, weight, Lipid profile, past history of angina, CKD, Migraine etc.
2. LDL/HDL ratio- it will be calculated from the lipid profile levels.
3. Insulin Resistance (HOMA IR)- According to Homeostatic Model Assessment of Insulin Resistance (HOMA IR) insulin resistance is calculated from serum insulin level and fasting glucose level.
4. hs CRP- It will be measured by ELISA
5. PANSS scale- Positive negative symptom scale for schizophrenia is used to measure the severity of positive symptoms, negative symptoms and general psychopathology in patients with schizophrenia.
6. CGI-SCH scale- Clinical Global Impression for schizophrenia is a scale that measures the baseline severity of illness, global improvement and the efficacy index.
7. Diet History Questionnaire - It is a 144-item questionnaire used in adults to know the diet history of a person over last 12 months. The scale has been used in order to standardize the diet of the participants between the study groups.

   Study design
   * The proposed study is a parallel arm, open label, randomized, controlled trial which will be conducted in patients with TRS on clozapine treatment for more than 6 months. The TRS patients on Clozapine, attending psychiatry OPD will be screened for metabolic syndrome using NCEP ATP III definition and those who are diagnosed as metabolic syndrome will be enrolled in the study. Out of the sample, 60 patients fulfilling the inclusion and exclusion criteria will be recruited for the study. The study will be conducted in the Department of Psychiatry, AIIMS, Bhubaneswar, over a period of 12 months. Written informed consent will be taken from the legally authorized representative (LAR) after explaining the objectives and procedure of the study in detail. The detailed history, relevant socio-demographic and clinical data will be collected in a structured case record form (CRF). At baseline, QRISK3 will be applied to measure the 10-year cardiovascular risk score. Serum Insulin level (for calculating insulin resistance), high sensitive C Reactive Protein (hs CRP) will be measured by ELISA technique. Fasting Plasma Glucose, and Lipid profile (Total Cholesterol, Triglyceride, LDL, HDL) level will be measured. In order to standardize the diet of all the participants, the investigators will use Diet History Questionnaire at the baseline which assess the diet of a person over last one year. PANSS and CGI-SCH will be administered to determine the baseline severity of illness.
   * The study sample will be randomized by computer-generated random numbers in 1:1 allocation ratio, with each group comprising of 30 patients. Group 1 will receive add-on Aripiprazole at a dose of 10 mg/day along with the ongoing clozapine and Metformin 500 mg twice a day treatment. The Group 2 will receive treatment as usual Metformin 500 mg twice a day along with ongoing Clozapine.
   * In the study population, PANSS, and CGI-SCH will be re-administered at the end of 3 months and 6 months, to evaluate the change in scores within each group and to compare the change between the two groups.
   * Diet History Questionnaire will be administered to all the participants after 6 months.
   * The QRISK 3, serum insulin, hs CRP, lipid profile, FBS will be administered at the baseline and at the end of 6 months in order to score the changes between the two groups.
   * The pre- and post-treatment rating using QRISK 3, PANSS, and CGI-SCH will be administered by a Psychiatrist, and the Serum insulin, CRP will be done by a pharmacologist. Both the outcome assessors will be blind to the treatment allocation.

   Study Duration - The study will be conducted for a period of 12 months. DETAILS OF INTERVENTIONS Standard of care The patients who are randomized to this group will receive the Clozapine in the usual dose along with Metformin 500mg twice a day.

   Add on aripiprazole The patients who are randomized to Aripiprazole group will receive Aripiprazole at a stable dose of 10 mg/day during the study period that is for 24 weeks along with Clozapine and Metformin 500 mg twice a day.
8. Statistical analysis:

   The continuous variables (serum insulin, serum hs CRP) will be presented as a mean and standard deviation and categorical data in percentage. Student t-test, the Paired t-test, ANOVA will be applied to parametric data and Mann-Whitney and Wilcoxon signed rank test will be applied for non-parametric data. For categorical data, Fischer's exact test will be used. Statistical software SPSS Version 22.0 will be used and p< 0.05 will be considered as statistically significant.

   Sample size calculation: Sample size calculation has been done on the basis of expected difference in cardiovascular risk scoring (QRISK3), which is the primary outcome measure of our study. Sample size of 23 per group can achieve a power of 80% to detect the difference of 5% in cardiovascular risk scoring (QRISK3) between the groups considering standard deviation as 6.0 and level of significance 0.05. Considering an attrition rate of 25%, 30 patients per group will be recruited.
9. Novelty/Innovation:

Metabolic syndrome is an emerging condition and it is more pronounced in TRS. Management of TRS is itself a challenging issue where the only option being Clozapine, it's use is further limited because of treatment emergent metabolic syndrome. There is limited option for the treatment of metabolic syndrome in TRS in the existing literature obtained from the various randomized placebo-controlled trials. The present study will be evaluating the efficacy and safety of Aripiprazole on the various metabolic parameters in TRS patients on Clozapine with metabolic syndrome.

10. Applicability/Relevance of the study:

1. If the outcome measures show a significant improvement with add on Aripiprazole, then add on Aripiprazole can be considered as a treatment option for metabolic syndrome in patients with TRS on clozapine.
2. Aripiprazole has been used as a successful augmenting agent with Clozapine in cases of TRS, hence a single agent will be effective in not only reducing metabolic syndrome but also reduction of symptom profile thereby reduces polypharmacy.
3. The addition of Aripiprazole can also reduce the dosage of clozapine for symptom control, thereby reducing other clozapine dose related adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* • Patients clinically diagnosed with TRS (TRRIP consensus criteria) on Clozapine for more than 6 months.

  * Patients with metabolic syndrome (NCEP ATP III Definition).
  * Patients aged above 25 years of either sex.
  * Patients/LAR giving voluntary written consent for participation in the study.

Exclusion Criteria:

* • Patient on combination of Clozapine with other antipsychotics.

  * Patients with any contraindication for Metformin/Aripiprazole.
  * History of psychoactive substance abuse or dependence.
  * Co-morbid psychiatric, major medical or neurological disorders.
  * History of organicity or significant head injury.
  * Pregnant and breastfeeding females.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in QRISK3 score (QRISK3 is an algorythm based software which calculates the score using various parameters. It is not an abbreviation.). | 6 months
  interpreted in terms of percentage. Score of more than 10 % would be considered as having risk of cardiovascular risk.

SECONDARY OUTCOMES:
Change in Low density lipoprotein (LDL)/High density lipoprotein (HDL) ratio. | 6 months
Change in Insulin Resistance. | 6 months
Change in Positive and negative symptom scale (PANSS) scores | 6 months
  It has positive, negative and general psychopathology scores witn each item score 0 to 7. Minimum score 30
Change in C reactive protein (CRP). | 6 months
Change in Clinical Global Improovement for Schizophrenia (CGI-SCH) scores | 6 months
  Clinical severity of illness and degree of improvement will be observed using this scale. the scoring will be from 0-7. 0=not assessed. 1=very much improved and 7= very much worse
Adverse events reported in both groups. | 6 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Saha S, Chant D, McGrath J. A systematic review of mortality in schizophrenia: is the differential mortality gap worsening over time? Arch Gen Psychiatry. 2007 Oct;64(10):1123-31. doi: 10.1001/archpsyc.64.10.1123. PMID 17909124
- [Result] Mitchell AJ, Vancampfort D, Sweers K, van Winkel R, Yu W, De Hert M. Prevalence of metabolic syndrome and metabolic abnormalities in schizophrenia and related disorders--a systematic review and meta-analysis. Schizophr Bull. 2013 Mar;39(2):306-18. doi: 10.1093/schbul/sbr148. Epub 2011 Dec 29. PMID 22207632
- [Result] Boden R, Edman G, Reutfors J, Ostenson CG, Osby U. A comparison of cardiovascular risk factors for ten antipsychotic drugs in clinical practice. Neuropsychiatr Dis Treat. 2013;9:371-7. doi: 10.2147/NDT.S40554. Epub 2013 Mar 19. PMID 23682213
- [Result] Zimbron J, Khandaker GM, Toschi C, Jones PB, Fernandez-Egea E. A systematic review and meta-analysis of randomised controlled trials of treatments for clozapine-induced obesity and metabolic syndrome. Eur Neuropsychopharmacol. 2016 Sep;26(9):1353-1365. doi: 10.1016/j.euroneuro.2016.07.010. Epub 2016 Aug 2. PMID 27496573
- [Result] Choi YJ. Efficacy of adjunctive treatments added to olanzapine or clozapine for weight control in patients with schizophrenia: a systematic review and meta-analysis. ScientificWorldJournal. 2015;2015:970730. doi: 10.1155/2015/970730. Epub 2015 Jan 13. PMID 25664341
- [Result] Bai YM, Lin CC, Chen JY, Chen TT, Su TP, Chou P. Association of weight gain and metabolic syndrome in patients taking clozapine: an 8-year cohort study. J Clin Psychiatry. 2011 Jun;72(6):751-6. doi: 10.4088/JCP.09m05402yel. Epub 2010 Nov 30. PMID 21208584